CLINICAL TRIAL: NCT04400058
Title: Efficacy and Safety of Octagam 10% Therapy in COVID-19 Patients With Severe Disease Progression
Brief Title: Octagam 10% Therapy in COVID-19 Patients With Severe Disease Progression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GAM10-10
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Octagam 10% (Experimental): Octagam 10%
  Interventions: Biological: Octagam 10%
- Saline Solution (Placebo Comparator): Placebo
  Interventions: Other: Saline Solution

INTERVENTIONS:
Biological: Octagam 10% — Octagam 10%, 2 g/kg divided by 4 days (0.5 g/kg/day), administered by intravenous infusion over approximately 2 hours per day over 4 consecutive days
  Arms: Octagam 10%
Other: Saline Solution — Placebo
  Arms: Saline Solution

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, Phase 3 study to evaluate if high-dose Octagam 10% therapy can stabilize or improve clinical status in patients with severe Coronavirus disease

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged ≥18years old
2. Provide voluntary, fully informed written and signed consent before any study-related procedures are conducted
3. Able to understand and comply with the relevant aspects of the study protocol
4. Laboratory (RT-PCR) confirmed COVID-19 infection on throat swab and/or sputum and/or lower respiratory tract samples
5. Hospitalized with a resting room-air SpO2 of ≤93% or PaO2/FiO2 ratio <300mmHg. Measurement can be taken from documented source records in the 24 hours prior to screening
6. Chest imaging confirming lung involvement

Exclusion Criteria:

1. Existence of other evidence that can explain pneumonia including but not limited to: Influenza A virus, influenza B virus, bacterial pneumonia (as suggested by the combined clinical picture, radiological findings and known laboratory results [eg, elevated procalcitonin >0.5ng/mL and concomitant neutrophilia]), known fungal pneumonia, suspected fungal pneumonia based on compromised immune system with a history of past fungal infections, noninfectious causes, etc.
2. Known history of serious allergic reactions, including anaphylaxis, to IVIG or its preparation components
3. Subjects with a history of thromboembolic event (TEE) within the last 12 months, such as deep vein thrombosis, pulmonary embolism, myocardial infarction, ischemic stroke, transient ischemic attack, peripheral artery disease (Fontaine IV)
4. Subjects with an underlying medical condition that can lead to hypercoagulable states and hyperviscosity such as antithrombin III deficiency, Factor V Leiden, Protein C deficiency, antiphospholipid syndrome and malignancy
5. Known history of selective IgA deficiency with antibodies against IgA
6. Subjects with conditions such as human immunodeficiency virus (HIV) infection, known acute or chronic hepatitis B or C (HBsAg positive or HCV ribonucleic acid (RNA) PCR positive or currently treated with antivirals), pulmonary fibrosis, elevated procalcitonin (> 0.5) with concomitant neutrophilia (elevated polys), heparin induced thrombocytopenia (HIT), and moderate to severe renal dysfunction (per investigator discretion based on estimated glomerular filtration rate [eGFR] <59 mL/min/1.73 m2, as defined by KDIGO Clinical Practice Guideline):

   * Moderately reduced GFR (G3a): GFR = 45 to 59 ml/min/1.73 m2
   * Moderately reduced GFR (G3b): GFR = 30 to 44 ml/min/1.73 m2
   * Severely reduced GFR (G4): GFR = 15 to 29 ml/min/1.73 m2
   * Kidney failure (G5): GFR <15 ml/min/1.73 m2
7. Currently requiring IMV (invasive mechanical ventilation or having received IMV during the last 30 days
8. Known clinically significant preexisting lung, heart, or neuromuscular disease that, in the investigator's opinion, would impact subject's ability to complete study or may confound the study results
9. Body weight >125 kg
10. Women who are pregnant or breast-feeding
11. Subjects who received COVID-19 convalescent plasma, IVIG products, anti-interleukin agents (eg, Tocilizumab), or interferons for their COVID-19 disease before enrollment or plan to receive this treatment during the course of the study
12. Enrolled in other experimental interventional studies or taking experimental medications (ie, convalescent plasma). Diagnostic studies can be allowed if the anticipated total blood volume to be drawn across both studies and for therapeutic purposes does not exceed 450 mL over any 8-week period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (14):
  - Octapharma Research Site, Sheffield, Alabama
  - Octapharma Research Site, Loma Linda, California
  - Octapharma Research Site, Newport Beach, California
  - Octapharma Research Site, Orange, California
  - Octapharma Research Site, San Diego, California
  - Octapharma Research Site, Washington D.C., District of Columbia
  - Octapharma Research Site, Honolulu, Hawaii
  - Octapharma Research Site, Iowa City, Iowa
  - Octapharma Research Site, Covington, Louisiana
  - Octapharma Research Site, Midland, Michigan
  - Octapharma Research Site, Las Vegas, Nevada
  - Octapharma Research Site, Minot, North Dakota
  - Octapharma Research Site, Charleston, South Carolina
  - Octapharma Research Site, Tyler, Texas
- Russia (3):
  - Octapharma Research Site, Ivanovo
  - Octapharma Research Site, Moscow
  - Octapharma Research Site, Ryazan
- Ukraine (3):
  - Octapharma Research Site, Ivano-Frankivsk
  - Octapharma Research Site, Kharkiv
  - Octapharma Research Site, Kremenchuk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 207 patients were enrolled between June 2020 and February 2021 at 23 sites across the United States, Russia and Ukraine
Groups:
- Saline Solution: Saline solution placebo group
Period: Overall Study
Arm/Group | Octagam 10% | Saline Solution
Started | 105 | 102
Completed | 84 | 86
Not Completed | 21 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octagam 10% | Saline Solution | Total
Number analyzed (Participants) | 105 | 102 | 207
Age, Continuous [Mean (Full Range); unit: years] | 57.6 [26 to 83] | 58.9 [30 to 89] | 58.2 [26 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 48 | 88
  Male | 65 | 54 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 21 | 41
  Not Hispanic or Latino | 73 | 76 | 149
  Unknown or Not Reported | 12 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 87 | 89 | 176
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 5 | 14
Body Mass Index (BMI)(kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 31.47 (5.570) | 32.33 (6.322) | 31.88 (5.934)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Reaching Stabilization or Improvement in Clinical Status at Day 7
Description: Proportion of subjects reaching stabilization or improvement in clinical status in at least one category on a 6-point clinical status scale.
  Clinical status categories will be defined as:
  1. Hospital discharge or meet discharge criteria (discharge criteria are defined as clinical recovery, i.e. no fever, respiratory rate, oxygen saturation return to normal, and cough relief).
  2. Hospitalization, not requiring supplemental oxygen.
  3. Hospitalization, requiring supplemental oxygen (but not NIV/HFNC).
  4. ICU/hospitalization, requiring NIV/HFNC therapy, as defined by A-a Gradient ≥150mmHg.
  5. ICU, requiring Extracorporeal Membrane Oxygenation (ECMO) and/or IMV.
  6. Death.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo
  Placebo: Placebo
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 105 | 102
Participants | 89 | 82

2. Secondary Outcome: Length of Hospital Stay (Time to Discharge)
Description: Median length of hospital stay in subjects treated with Octagam 10%, compared to those that received placebo from randomization through Day 33
Time Frame: 33 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 105 | 102
days | 12 [9 to 14] | 11 [9 to 15]

3. Secondary Outcome: Number of Subjects Reaching Stabilization or Improvement In Clinical Status at Day 14
Description: Number of subjects with maintenance or improvement by at least one category on the 6-point clinical status scale on Day 14.
  Clinical status categories will be defined as:
  1. Hospital discharge or meet discharge criteria (discharge criteria are defined as clinical recovery, i.e. no fever, respiratory rate, oxygen saturation return to normal, and cough relief).
  2. Hospitalization, not requiring supplemental oxygen.
  3. Hospitalization, requiring supplemental oxygen (but not NIV/HFNC).
  4. ICU/hospitalization, requiring NIV/HFNC therapy, as defined by A-a Gradient ≥ 150 mmHg.
  5. ICU, requiring Extracorporeal Membrane Oxygenation (ECMO) and/or IMV.
  6. Death.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 105 | 102
Participants | 86 | 83

4. Secondary Outcome: Cumulative Duration of Invasive Mechanical Venitlation (IMV)
Description: Duration of invasive mechanical ventilation in subjects treated with Octagam 10% compared to placebo from randomization through Day 33
Time Frame: 33 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 105 | 102
days | 2.7 (8.05) | 1.6 (5.95)

5. Secondary Outcome: Number of Subjects With Severe Disease Progression
Description: Number of subjects who experienced severe disease progression while treated with Octagam 10% compared to those that received placebo at Day 33. Severe disease progression is defined as subjects requiring extracorporeal membrane oxygenation, mechanical ventilation and/or died through day 33.
Time Frame: 33 days
Measure: Count of Participants; unit: Participants
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 105 | 102
Participants | 15 | 12

6. Secondary Outcome: ICU Stay Length
Description: Average length of ICU stay in subjects treated with Octagam 10% compared to those that received placebo from randomization through Day 33.
Time Frame: 33 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 105 | 102
days | 4.6 (10.08) | 3.9 (8.83)

7. Secondary Outcome: Cumulative Mortality Rate Through Day 33
Description: Cumulative mortality in subjects treated with Octagam 10% compared to those that received placebo at Day 33
Time Frame: 33 days
Measure: Count of Participants; unit: Participants
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 105 | 102
Participants | 12 | 6

8. Post Hoc Outcome: Post Study Health Status, Any Residual Health Effects From COVID-19 or the Study Treatment - 3 Months Post-Study (COVID-19 Subject Questionnaire)
Description: Subjects who completed the core study and entered the registry were administered questionnaires at 3 months asking about their general health. Subjects were asked:
  How is your general health?
  1. Poor
  2. Fair
  3. Good
  4. Very Good
  5. Excellent
  6. Missing
  How would you compare your general health now to what it was before you were ill with Covid-19?
  1. Much worse
  2. Somewhat worse
  3. The same
  4. Somewhat better
  5. Much better
  6. Missing
  Since last contact, have you?
  1. Been hospitalized
  2. Sought consultation from a health care professional
  3. Experienced deterioration of your health without seeking HCP consultation
  4. None of the above
  5. Missing
  If the above question was not "none of the above", was it in relation to the symptoms?
  1. Other
  2. Similar to the symptoms experienced during COVID-19 hospitalization
  Prior to Covid-19 did you work or go to school full time?
  1. Yes
  2. No
  Do you currently work or go to school full time?
  1. Yes
  2. No
Time Frame: 3 months post-study
Measure: Number; unit: participants
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 84 | 84
participants
  Question 1 - Poor | 1 | 1
  Question 1 - Fair | 14 | 24
  Question 1 - Good | 30 | 30
  Question 1 - Very Good | 19 | 15
  Question 1 - Excellent | 6 | 5
  Question 1 - Missing Answer | 14 | 9
  Question 2 - Much Worse | 3 | 5
  Question 2 - Somewhat Worse | 18 | 29
  Question 2 - The Same | 29 | 29
  Question 2 - Somewhat Better | 11 | 7
  Question 2 - Much Better | 9 | 5
  Question 2 - Missing Answer | 14 | 9
  Question 3 - Been Hospitalized | 2 | 7
  Question 3 - Sought consultation from HCP | 21 | 25
  Question 3 - Experienced deterioration of your health without HCP documentation | 4 | 8
  Question 3 - None of the above | 43 | 38
  Question 3 - Missing answer | 14 | 9
  Question 4 - Other | 23 | 27
  Question 4 - Similar to those during the COVID-19 hospitalization | 9 | 13
  Question 5 - Yes | 53 | 49
  Question 5 - No | 17 | 26
  Question 6 - Yes | 45 | 42
  Question 6 - No | 25 | 32

9. Post Hoc Outcome: Post Study Health Status, Any Residual Health Effects From COVID-19 or the Study Treatment - 6 Months Post-Study (COVID-19 Subject Questionnaire)
Description: Subjects who completed the core study and entered the registry were administered questionnaires at 6 months asking about their general health. Subjects were asked:
  How is your general health?
  1. Poor
  2. Fair
  3. Good
  4. Very Good
  5. Excellent
  6. Missing
  How would you compare your general health now to what it was before you were ill with Covid-19?
  1. Much worse
  2. Somewhat worse
  3. The same
  4. Somewhat better
  5. Much better
  6. Missing
  Since last contact, have you?
  1. Been hospitalized
  2. Sought consultation from a health care professional
  3. Experienced deterioration of your health without seeking HCP consultation
  4. None of the above
  5. Missing
  If the above question was not "none of the above", was it in relation to the symptoms?
  1. Other
  2. Similar to the symptoms experienced during COVID-19 hospitalization
  Prior to Covid-19 did you work or go to school full time?
  1. Yes
  2. No
  Do you currently work or go to school full time?
  1. Yes
  2. No
Time Frame: 6 months post-study
Measure: Number; unit: participants
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 84 | 84
participants
  Question 1 - Poor | 0 | 0
  Question 1 - Fair | 15 | 20
  Question 1 - Good | 26 | 22
  Question 1 - Very Good | 18 | 19
  Question 1 - Excellent | 4 | 7
  Question 1 - Missing Answer | 21 | 16
  Question 2 - Much Worse | 3 | 4
  Question 2 - Somewhat Worse | 12 | 12
  Question 2 - The Same | 30 | 38
  Question 2 - Somewhat Better | 8 | 9
  Question 2 - Much Better | 10 | 5
  Question 2 - Missing Answer | 21 | 16
  Question 3 - Been Hospitalized | 0 | 3
  Question 3 - Sought consultation from HCP | 12 | 16
  Question 3 - Experienced deterioration of your health without HCP documentation | 1 | 0
  Question 3 - None of the above | 49 | 49
  Question 3 - Missing answer | 22 | 16
  Question 4 - Other | 6 | 18
  Question 4 - Similar to those during the COVID-19 hospitalization | 6 | 4
  Question 5 - Yes | 49 | 43
  Question 5 - No | 13 | 25
  Question 6 - Yes | 41 | 39
  Question 6 - No | 21 | 29

10. Post Hoc Outcome: Post Study Health Status, Any Residual Health Effects From COVID-19 or the Study Treatment - 9 Months Post-Study (COVID-19 Subject Questionnaire)
Description: Subjects who completed the core study and entered the registry were administered questionnaires at 9 months asking about their general health. Subjects were asked:
  How is your general health?
  1. Poor
  2. Fair
  3. Good
  4. Very Good
  5. Excellent
  6. Missing
  How would you compare your general health now to what it was before you were ill with Covid-19?
  1. Much worse
  2. Somewhat worse
  3. The same
  4. Somewhat better
  5. Much better
  6. Missing
  Since last contact, have you?
  1. Been hospitalized
  2. Sought consultation from a health care professional
  3. Experienced deterioration of your health without seeking HCP consultation
  4. None of the above
  5. Missing
  If the above question was not "none of the above", was it in relation to the symptoms?
  1. Other
  2. Similar to the symptoms experienced during COVID-19 hospitalization
  Prior to Covid-19 did you work or go to school full time?
  1. Yes
  2. No
  Do you currently work or go to school full time?
  1. Yes
  2. No
Time Frame: 9 months post-study
Measure: Number; unit: participants
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 84 | 84
participants
  Question 1 - Poor | 1 | 1
  Question 1 - Fair | 10 | 19
  Question 1 - Good | 29 | 31
  Question 1 - Very Good | 19 | 14
  Question 1 - Excellent | 4 | 4
  Question 1 - Missing Answer | 21 | 15
  Question 2 - Much Worse | 3 | 4
  Question 2 - Somewhat Worse | 13 | 15
  Question 2 - The Same | 28 | 38
  Question 2 - Somewhat Better | 10 | 6
  Question 2 - Much Better | 9 | 6
  Question 2 - Missing Answer | 21 | 15
  Question 3 - Been Hospitalized | 0 | 2
  Question 3 - Sought consultation from HCP | 17 | 24
  Question 3 - Experienced deterioration of your health without HCP documentation | 5 | 1
  Question 3 - None of the above | 41 | 43
  Question 3 - Missing answer | 21 | 15
  Question 4 - Other | 15 | 23
  Question 4 - Similar to those during the COVID-19 hospitalization | 9 | 4
  Question 5 - Yes | 49 | 44
  Question 5 - No | 14 | 25
  Question 6 - Yes | 46 | 44
  Question 6 - No | 17 | 25

11. Post Hoc Outcome: Post Study Health Status, Any Residual Health Effects From COVID-19 or the Study Treatment - 1 Year Post-Study (COVID-19 Subject Questionnaire)
Description: Subjects who completed the core study and entered the registry were administered questionnaires at 1 year asking about their general health. Subjects were asked:
  How is your general health?
  1. Poor
  2. Fair
  3. Good
  4. Very Good
  5. Excellent
  6. Missing
  How would you compare your general health now to what it was before you were ill with Covid-19?
  1. Much worse
  2. Somewhat worse
  3. The same
  4. Somewhat better
  5. Much better
  6. Missing
  Since last contact, have you?
  1. Been hospitalized
  2. Sought consultation from a health care professional
  3. Experienced deterioration of your health without seeking HCP consultation
  4. None of the above
  5. Missing
  If the above question was not "none of the above", was it in relation to the symptoms?
  1. Other
  2. Similar to the symptoms experienced during COVID-19 hospitalization
  Prior to Covid-19 did you work or go to school full time?
  1. Yes
  2. No
  Do you currently work or go to school full time?
  1. Yes
  2. No
Time Frame: 1-year post-study
Measure: Number; unit: participants
Arm/Group | Octagam 10% | Placebo
Number analyzed (Participants) | 84 | 84
participants
  Question 1 - Poor | 1 | 1
  Question 1 - Fair | 11 | 14
  Question 1 - Good | 35 | 36
  Question 1 - Very Good | 17 | 13
  Question 1 - Excellent | 2 | 3
  Question 1 - Missing Answer | 18 | 17
  Question 2 - Much Worse | 2 | 3
  Question 2 - Somewhat Worse | 15 | 12
  Question 2 - The Same | 32 | 44
  Question 2 - Somewhat Better | 12 | 5
  Question 2 - Much Better | 5 | 3
  Question 2 - Missing Answer | 18 | 17
  Question 3 - Been Hospitalized | 1 | 2
  Question 3 - Sought consultation from HCP | 29 | 22
  Question 3 - Experienced deterioration of your health without HCP documentation | 2 | 0
  Question 3 - None of the above | 34 | 43
  Question 3 - Missing answer | 18 | 17
  Question 4 - Other | 27 | 21
  Question 4 - Similar to those during the COVID-19 hospitalization | 5 | 5
  Question 5 - Yes | 50 | 44
  Question 5 - No | 16 | 23
  Question 6 - Yes | 44 | 44
  Question 6 - No | 22 | 23

ADVERSE EVENTS:
Time Frame: 33 days
Description: Safety Population (SAF) analysed. SAF includes all subjects who are randomized and received any amount of IVIG or placebo. The analysis was conducted according to the treatment which subjects actually received.
Arm/Group | Octagam 10% | Placebo
All-Cause Mortality (participants affected / at risk) | 13/105 | 6/102
Serious Adverse Events (participants affected / at risk) | 15/105 | 12/100
Other Adverse Events (participants affected / at risk) | 49/105 | 40/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octagam 10% (N=105) | Placebo (N=100)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 3 (3)
COVID-19 Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Viral Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Viral Cardiomyopathy (Infections and infestations) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary Failure (Cardiac disorders) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 3 (3) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic Hyperglycaemic Coma (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octagam 10% (N=105) | Placebo (N=100)
Constipation (Gastrointestinal disorders) | 10 (10) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Anxiety (Psychiatric disorders) | 8 (8) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (7) | 5 (5)
Headache (Nervous system disorders) | 10 (10) | 7 (7)
Acute Kidney Injury (Renal and urinary disorders) | 7 (7) | 5 (5)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)

LIMITATIONS AND CAVEATS:
Post-hoc outcomes were recorded for subjects who chose to enter the post-study phone call registry, therefore, the numbers differ from the overall study population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04400058/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT04400058/SAP_001.pdf